CLINICAL TRIAL: NCT04585113
Title: Diagnostic Value of Dual-energy CT to Detect and Characterize Crystal Deposits in Patients With Hand Osteoarthritis Undergoing Hand Surgery: a Diagnostic Accuracy Study
Brief Title: Diagnostic Accuracy of Dual-energy CT
Acronym: DAD
Status: Completed | Type: Observational
Sponsor: Henning Bliddal (Other)
Responsible Party: Sponsor-Investigator, Henning Bliddal, MD, DMSci, Professor of Rheumatology, Frederiksberg University Hospital
Organization: Frederiksberg University Hospital (Other)
Other Study IDs: DAD2020
Record Dates: First submitted 2020-09-30; First posted 2020-10-14 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Osteoarthritis; Hand Osteoarthritis; Crystal; Deposit Joint; Crystals; Arthritis, Pyrophosphate; Crystals; Arthritis, Hydroxyapatite; Crystal Arthritis; Crystal Arthropathy of Hand
MeSH Terms: conditions — Osteoarthritis; Arthritis; Crystal Arthropathies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Material obtained during surgery from the joint.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People with hand OA awaiting surgery: Patients with hand OA awaiting hand surgery of a joint with OA will be considered eligible. All IP joints in the hands are eligible (thus both IP, PIP and DIP) if in- and exclusion criteria are fulfilled.
  Interventions: Radiation: CT-scanning

INTERVENTIONS:
Radiation: CT-scanning — All participants will receive dual-energy CT scanning and cone-beam CT scanning prior surgery.

SUMMARY:
The study will include 20 people with hand OA awaiting surgery in the fingers. Participants will undergo dual-energy CT, cone-beam CT, ultrasound, clinical examination, blood sampling and questionnaires. Images will be analysed for the presence of joint-associated crystal including monosodium urate, calcium pyrophosphate and calcium hydroxyapatite. Material obtained during surgery will be used for crystal verification and calculation of diagnostic accuracy of dual-energy CT and cone-beam CT.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Informed consent obtained.
3. Patients with hand OA as defined by the American College of Rheumatology Classification Criteria for hand OA:

   * Hand pain, aching or stiffness

And 3 or 4 of the following features:

* Hard tissue enlargement of ≥2 of the 10 selected joints*.
* Hard tissue enlargement of ≥2 of the 10 DIP joints.
* Fewer than 3 swollen MCP joints.
* Deformity of at least 1 of 10 selected joints*. *The 10 selected joints are the second and third DIP, the second and third PIP, and the first carpometacarpal joints of both hands.

Exclusion Criteria:

1. Known inflammatory rheumatic diseases (e.g. rheumatoid arthritis, gout, psoriatic arthritis, psoriasis, inflammatory bowel disease), or other joint diseases (haemochromatosis)
2. Positive anti-cyclic citrullinated peptide (>10 kU/L)
3. Known cutaneous deposition diseases (e.g. amyloidosis or porphyria).
4. Foreign material/metallic implants at the area of interest will be excluded to avoid artefacts on CBCT [68].
5. Other diseases in the area - e.g. skin disease, known previous fracture in the joint of interest.
6. Participation in experimental device or experimental drug study 3 months prior to enrolment.
7. Pregnancy or breast-feeding.
8. Previous septic arthritis at the target joint.
9. Previous surgical procedures at the target joint.
10. Injection into the target joint within 3 months prior to enrolment.
11. Inability to speak and read Danish fluently.
12. Treatment with Colchicine within the last 30 days.
13. Treatment with systemic steroids ≥7.5 mg prednisolone within the last 30 days.
14. Lack of sample obtained for reference standard, i.e. unable to obtain either synovial fluid, joint lavage fluid, joint biopsy or excite joint.
15. Any other condition that in the opinion of the investigator may interfere with study participation.

There will be no restriction on sex or Kellgren-Lawrence (KL) grading.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hand OA awaiting hand surgery of a joint with OA will be considered eligible.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
Positive likelihood ratio | 20 months
  To determine the positive likelihood ratio of DECT to detect crystal deposition in an osteoarthritic joint of the hand.
Discriminating joint-associated crystals | 20 months
  To determine DECTs ability to discriminate MSU from calcium-containing crystals in an osteoarthritic joint of the hand.

SECONDARY OUTCOMES:
Negative likelihood ratio | 20 months
  To determine the negative likelihood ratio of DECT to detect crystal deposition in an osteoarthritic joint of the hand.
Inflammation | 20 months
  Synovitis-score of inflammation detected by ultrasound
Relationship between inflammation and crystals | 20 months
  Analysis of covariance (ANCOVA), with a factor for presence of crystals (X=1 or X=0), and synovitis score as dependent variable.
Degenerative status | 20 months
  Described by KL-score
Relationship between KL-score and crystals | 20 months
  Analysis of covariance (ANCOVA), with a factor for presence of crystals (X=1 or X=0), and KL-score as dependent variable.
Erosions score | 20 months
  Erosions as estimated by the hand osteoarthritis magnetic resonance imaging scoring system (HOAMRIS) for erosions evaluated by CBCT
Relationship between erosion-score and crystals | 20 months
  Analysis of covariance (ANCOVA), with a factor for presence of crystals (X=1 or X=0), and erosion-score as dependent variable.

CONTACTS AND LOCATIONS:
Overall Officials: Henning Bliddal, MD, DMSc, Principal Investigator — Parker Instituttet
Locations (1):
- The Parker Institute, Bispebjerg and Frederiksberg Hospital, Copenhagen, DK, Denmark

IPD SHARING:
Plan to Share IPD: Undecided